CLINICAL TRIAL: NCT01280240
Title: Open-label Pharmacokinetic Study of Iron Isomaltoside 1000 (Monofer®) Administered by 250 mg IV Bolus Injection or 500 mg Intravenous Infusion to Patients With Non-hematological Malignancies Associated With Chemotherapy Induced Anaemia (CIA).
Brief Title: Pharmacokinetic Study of Iron Isomaltoside 1000 Administered by 250 mg IV Bolus Injection or 500 mg Intravenous Infusion to Patients With Non-hematological Malignancies Associated With Chemotherapy Induced Anaemia
Acronym: PK-CIA-06
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmacosmos A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: P-Monofer-PK-CIA-06; PK-CIA-06
Record Dates: First submitted 2011-01-19; First posted 2011-01-20 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Patients With Chemotherapy Induced Anemia (CIA)
Keywords: anemia; cancer; CIA
MeSH Terms: conditions — Anemia; Neoplasms | interventions — iron isomaltoside 1000

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Monofer 500 mg (Active Comparator)
  Interventions: Drug: Monofer(R)
- Monofer 250 mg (Active Comparator)
  Interventions: Drug: Monofer(R)

INTERVENTIONS:
Drug: Monofer(R) — Intravenous bolus injection given over app. 2 minutes only once
  Other Names: iron isomaltoside 1000

SUMMARY:
The purpose of this study is to assess Pharmakokinetic properties of iron isomaltoside 1000 (Monofer®) in doses of 250 mg and 500 mg in patients suffering from Chemotherapy Induced anemia.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged more than 18 years.
2. Weight above 50 kg.
3. Subjects diagnosed with non-hematological malignancies (solid tumors only) receiving chemotherapy at least 1 day prior to screening and who are going to receive at least two more chemotherapy cycles.
4. Hb < 12 g/dL.
5. TfS <20%.
6. Serum Ferritin <800 ng/ml.
7. An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
8. Willingness to participate after informed consent.

Exclusion Criteria:

1. Anaemia caused primarily by other factors than CIA.
2. IV or oral iron treatment within 4 weeks prior to screening visit.
3. Erythropoietin treatment within 4 weeks prior to screening visit.
4. Blood transfusion within 4 weeks prior to screening visit.
5. Imminent expectation of blood transfusion on part of treating physician.
6. Iron overload or disturbances in utilization of iron (e.g. haemochromatosis and haemosiderosis).
7. Drug hypersensitivity (i.e. previous hypersensitivity to Iron Dextran or iron mono- or disaccharide complexes).
8. Known hypersensitivity to any excipients in the investigational drug products.
9. Subjects with a history of multiple allergies.
10. Decompensated liver cirrhosis and hepatitis (alanine aminotransferase (ALAT) > 3 times upper normal limit).
11. History of Immunocompromise and/or history of Hepatitis B and/or C.
12. Active acute or chronic infections (assessed by clinical judgement and if deemed necessary by investigator supplied with white blood cells (WBC) and C-reactive protein (CRP)).
13. Rheumatoid arthritis with symptoms or signs of active joint inflammation.
14. Pregnant or breast feeding women.
15. Women of child bearing potential who are not using safe contraceptive methods (e.g. intrauterine device, oral contraceptives or surgically sterilized) or who are planning to become pregnant within the study period.
16. Planned elective surgery during the study.
17. Participation in any other clinical study (except chemotherapy protocol) within 3 months prior to screening.
18. Untreated B12 or folate deficiency.
19. Any other medical condition that, in the opinion of Principal Investigator, may cause the subject to be unsuitable for the completion of the study or place the subject at potential risk from being in the study. Example, Uncontrolled Hypertension, Unstable Ischemic Heart Disease or Uncontrolled Diabetes Mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-03; Primary Completion 2012-09 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Total serum iron pharmacokinetic parameters: AUC0-t, AUC Cmax, Tmax, Ke, and T1/2 estimated from plasma/serum concentration profile from exposure to 7 days post-exposure. | 0-7 days

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Baltimore, MD, Maryland
  - Gabrail Cancer Center, Canton, Ohio